CLINICAL TRIAL: NCT00181558
Title: Atrasentan and Zometa for Men With Androgen Independent Prostate Cancer Metastatic to Bone: A Randomized Pilot Study
Brief Title: Atrasentan and Zometa for Men With Prostate Cancer Metastatic to Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Abbott (Industry)
Responsible Party: Matthew R. Smith, MD, PhD, Massachusetts General Hospital, Boston, MA 02114
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-200
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: Prostate Cancer; bone metastases; Atrasentan; Zometa; Androgen Independent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atrasentan; Zoledronic Acid

INTERVENTIONS:
Drug: Atrasentan
Drug: Zoledronic Acid (Zometa)

SUMMARY:
The main purpose of this study is to look at the effects (good or bad) that Atrasentan given alone and Atrasentan given with Zometa has on levels of bone formation and bone destruction in men with prostate cancer that has spread to the bones.

DETAILED DESCRIPTION:
* Patients will be randomized to either receive Atrasentan alone or Atrasentan plus Zometa.
* Patients receiving Atrasentan alone will receive this drug in pill form once daily for 12 weeks. Patients will have a physical exam, blood work, and a urine sample performed once every other week during the first four weeks of medication administration. After those two initial visits, they will return to the clinic once every 4 weeks to have the same tests repeated. A bone scan and abdominal-pelvic CT Scan will be done every 12 weeks.
* After the patient has been taking Atrasentan for 12 weeks, if the disease has not progressed, they will begin combination treatment of Atrasentan and Zometa.
* Patients receiving Atrasentan plus Zometa, receive Zometa intravenously and then immediately start Atrasentan orally once daily as long as they remain on the study. Patients will return to the clinic twice over the first 4 weeks (once every other week) to have a physical exam, blood work and urine test performed. After these two initial visits, they will return to the clinic once every 4 weeks to have the tests repeated and to receive another treatment of zometa. A bone scan and an abdominal-pelvic CT Scan will be done once every 12 weeks.
* Patients participation in this study will last as long as the disease does not progress and they are not experiencing any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* History of bilateral orchiectomy or current treatment with a GnRH agonist or antagonist
* Radiographically documented bone metastases
* Disease progression according to criteria from the PSA Working Group

Exclusion Criteria:

* Prior treatment with Atrasentan or Zometa within one year
* Serum creatinine > 2.0mg/dL
* Documented cardiovascular disability status of New York Heart Association Class 2
* Treatment with chemotherapy, radiation, steroids, estrogens, or PC-SPES within 6 weeks
* Treatment with bisphosphonates or radiopharmaceuticals within 12 weeks
* History of Paget's disease, hyperthyroidism, hyperparathyroidism, Cushing's syndrome, hyperprolactinemia or other disorder associated with metabolic bone disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2001-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To compare the effects of Atrasentan monotherapy with combination therapy using Atrasentan and Zometa on bone specific alkaline phosphatase.

SECONDARY OUTCOMES:
To evaluate the effects of Atrasentan monotherapy and combination therapy with Atrasentan and Zometa on PSA doubling time.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906